CLINICAL TRIAL: NCT04638608
Title: A Complex Intervention Study on a Palliative Rehabilitation Blended Learning Program to Support Relatives and Health Care Providers of People With ALS and FTD in Coping With Challenges
Brief Title: A Complex Intervention Study on a Palliative Rehabilitation Blended Learning Program to Support Relatives and Health Care Providers of People With ALS and Cognitive Impairments in Coping With Challenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Rehabilitation Centre for Neuromuscular Diseases (Other)
Responsible Party: Principal Investigator, Lene Klem Olesen, PhD, Occupational Therapist, MA in Educational psychology, Danish Rehabilitation Centre for Neuromuscular Diseases
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: DanishRebCND
Record Dates: First submitted 2020-11-10; First posted 2020-11-20 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Relatives; Health Care Providers; Cognitive Impairment; Rehabilitation
Keywords: Relatives, informal carer, family carer; ALS/MND; Cognitive impairment; Palliative rehabilitation; Blended learning; Online support, telehealth, e-learning; Peer-support; Health care providers
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Health Personnel

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMBRACE (Relatives) (Other): Feasibility test of a new palliative rehabilitation blended learning program for relatives of people with ALS/cognitive impairments
  Interventions: Other: EMBRACE (relatives)
- EMBRACE (Health care providers) (Other): Feasibility test of a new palliative rehabilitation blended learning program health care providers helping people with ALS/cognitive impairments
  Interventions: Other: EMBRACE (Health care providers)

INTERVENTIONS:
Other: EMBRACE (relatives) — Online support program for both relatives
  Arms: EMBRACE (Relatives)
Other: EMBRACE (Health care providers) — Online support program for health care providers
  Arms: EMBRACE (Health care providers)

SUMMARY:
A complex intervention study on a palliative rehabilitation blended learning program to support relatives and health care providers of people with ALS and cognitive impairments in coping with challenges.

DETAILED DESCRIPTION:
The projects concerns tree studies.

1. Identifying experience-based evidence of relative of deceased people with ALS/cognitive impairments and health care providers (working with these persons) and develop an intervention program.
2. Developing a palliative rehabilitation blended learning program for relatives of people with ALS and cognitive impairments and for the health care providers.
3. Feasibility testing of the two palliative rehabilitation blended learning programs for relatives and health care providers.

Though online palliative rehabilitation the intervention aims to support both relatives of people with ALS/cognitive impairments and health care providers in coping with challenges related to the diseases.

The intervention consists of blended learning through online videos and virtual group meetings, where peer-support play an essential role. The videos consists of a psycho education, mindfulness based stress reduction, relationship changes, intimacy, sorrow and grief, control management, planning the future, how to communicate, hope, creating memories, external support offers. Besides the videos and group meetings, the relatives are given the possibility to make Ecomaps and diary reflections.

ELIGIBILITY:
Inclusion Criteria: Relatives

* relatives (spouse or partner) living with a person with ALS and cognitive impairments (rated on the ALS-FTD-Q by the relative, cut-off >22) Able to talk and understand proficient danish referred to the national rehabilitation center for neuromuscular diseases and have had a visit from an als-consultant

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Coping with ALS and cognitive impairments | 0-4 month
  Framework of Complex Intervention in Health: MRC-guidelines according to acceptability, implementation and integration

SECONDARY OUTCOMES:
Burden | 0-4 month
  The Zarit Burden Interview (ZBI-22) questionnaires at baseline (Pre and post intervention)
Anxiety and Stress | 0-4 month
  Hospital Anxiety and Depression Scale (HADS) (Pre and post intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Handberg, senior researcher, Study Chair — The National Rehabilitation Center for Neuromuscular Diseases
Locations (1):
- The Danish national Rehabilitation Center for neuromuscular diseases, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olesen LK, la Cour K, Nimmon L, With H, Handberg C. Experiences of an Online Palliative Rehabilitation Programme for Spousal Caregivers of People With Amyotrophic Lateral Sclerosis and Cognitive and/or Behavioural Impairments: A Qualitative Interpretive Study. Adv Rehabil Sci Pract. 2024 Feb 9;13:27536351241227860. doi: 10.1177/27536351241227860. eCollection 2024 Jan-Dec. PMID 38343431
- [Derived] Olesen LK, la Cour K, With H, Mahoney AF, Handberg C. A cross-sectional evaluation of acceptability of an online palliative rehabilitation program for family caregivers of people with amyotrophic lateral sclerosis and cognitive and behavioral impairments. BMC Health Serv Res. 2022 May 24;22(1):697. doi: 10.1186/s12913-022-07986-4. PMID 35610609
- [Derived] Olesen LK, la Cour K, With H, Handberg C. Reflections of family caregivers and health professionals on the everyday challenges of caring for persons with amyotrophic lateral sclerosis and cognitive impairments: a qualitative study. Palliat Care Soc Pract. 2022 Feb 15;16:26323524221077702. doi: 10.1177/26323524221077702. eCollection 2022. PMID 35187490